CLINICAL TRIAL: NCT04955964
Title: Post Authorization Study to Monitor Efficacy, Effectiveness and Safety of Lanadelumab (Takhzyro®) in Patients Aged 12 Years and Older With Hereditary Angioedema (HAE) in Argentina
Brief Title: A Study of Lanadelumab in Teenagers and Adults With Hereditary Angioedema (HAE) in Argentina
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4008
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Angioedemas, Hereditary
Keywords: Lanadelumab; Post-authorization study
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with diagnosis of HAE who have received at least one dose of lanadelumab according to currently approved indications in routine clinical practice settings in Argentina will be observed in this study.

SUMMARY:
The main aim of this study is to learn about the safety profile of lanadelumab in teenagers and adults with hereditary angioedema (HAE) in Argentina as part of routine routine practice.

This study is about collecting data only. The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study. The study will collect data from the participant's medical records.

Participants do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants (>=12 years) with investigator confirmed diagnosis of HAE.
* Have received at least one dose of lanadelumab according to approved indications.
* Signed the mandatory consent that has been agreed with national regulatory authorities (ANMAT) as applicable.

Exclusion Criteria:

- Hypersensitivity to the active substance or to any of the excipients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will include all participants treated with lanadelumab according to approved indications in routine clinical practice settings in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Baseline up to end of study (up to 24 months)
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Percentage of participants with AESIs such as hypersensitivity, immunogenicity, liver toxicity, and embryo-fetal toxicity will be reported.
Percentage of Participants With Serious and Non-serious Adverse Events (AEs) | Baseline up to end of study (up to 24 months)
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Serious AE is any untoward medical occurrence (whether considered to be related to study assigned treatment or not) that at any dose resulted in death, is life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital abnormality/birth defect, or was an important medical event. AEs including both serious and non-serious adverse events will be reported.

SECONDARY OUTCOMES:
Monthly Mean Rate of Investigator Confirmed HAE Attacks | At Weeks 12 and 24
  HAE attack is defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema based on investigator judgement. In general, the event must have symptoms or signs consistent with an attack in greater than or equal to (>=) 1 of the typical locations (peripheral angioedema; abdominal angioedema; laryngeal/tongue angioedema). Monthly mean rate of investigator confirmed HAE attacks with assessments at Weeks 12 and 24 will be reported.
Monthly Mean Rate of Investigator Confirmed Moderate or Severe HAE Attacks | At Weeks 12 and 24
  The overall severity of attack will be determined by the investigator using following definitions: mild (transient or mild discomfort), moderate (mild to moderate limitation in activity), severe (marked limitation in activity). Monthly mean rate of investigator confirmed moderate or severe HAE attacks with assessments at Weeks 12 and 24 will be reported.
Monthly Mean Rate of Investigator Confirmed HAE Attacks Requiring Acute Treatment | At Weeks 12 and 24
  HAE attack is defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema based on investigator judgement. In general, the event must have symptoms or signs consistent with an attack in >=1 of the typical locations (peripheral angioedema; abdominal angioedema; laryngeal/tongue angioedema). Monthly mean rate of investigator confirmed HAE attacks requiring acute treatment with assessments at Weeks 12 and 24 will be reported.
Percentage of Participants who are Attack Free | At Weeks 12 and 24
  A participant will be considered as attack free during an efficacy evaluation period if the participant has no investigator-confirmed HAE attacks during treatment period. HAE attack is defined as a discrete episode during which the participant progressed from no angioedema to symptoms of angioedema based on investigator judgement. In general, the event must have symptoms or signs consistent with an attack in >=1 of the typical locations (peripheral angioedema; abdominal angioedema; laryngeal/tongue angioedema). Percentage of participants who are attack free with assessments at 12 and 24 weeks will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Ic Projects Srl, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60e84e971f1122001e30a94f